CLINICAL TRIAL: NCT02276300
Title: A Phase 1 Study of Peptide Vaccination for the Treatment of Patients With Solid Tumors Moderately Expressing HER2/Neu
Brief Title: HER2-Peptide Vaccination of Patients With Solid Tumors
Acronym: HER2
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Technical University of Munich (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ATZ-1068-KRA-20I
Record Dates: First submitted 2014-09-25; First posted 2014-10-28 (Estimated); Last update posted 2019-11-20 (Actual); Status verified 2019-11

CONDITIONS: Gastric Cancer; Breast Cancer
MeSH Terms: conditions — Stomach Neoplasms; Breast Neoplasms | interventions — Cyclophosphamide; sargramostim; Imiquimod

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- HER2-Peptid-Vakzine, Cyclophosphamide (Experimental): Her2-peptide vaccination, Sargramostim, Imiquimod, Cyclophosphamide
  Interventions: Drug: Cyclophosphamide; Drug: Sargramostim; Drug: HER2-Peptid-Vakzine; Drug: Imiquimod

INTERVENTIONS:
Drug: Cyclophosphamide — Treatment of mild Endoxan application three days before Her2 vaccination
  Other Names: Endoxan
Drug: Sargramostim — Sargramostim is part of Her2 vaccination
  Other Names: Leukine
Drug: HER2-Peptid-Vakzine — Her2 vaccination is supplemented by Sargramostim and Aldara Creme application
Drug: Imiquimod — Imiquimod is part of Her2 vaccination
  Other Names: Aldara 5% Crème

SUMMARY:
Investigation of peptide vaccination targeting HER2/neu in patients with metastasized breast or gastric cancer with moderate HER2/neu expression.

DETAILED DESCRIPTION:
This is an interventional phase I clinical study to investigate the safety, tolerability and efficacy of HER2-derived peptide vaccination. HLA-A2+ patients with stage IV metastasized breast or gastric cancer with HER2 expression (IHC Score 2+) without gene amplification proved by FISH analysis, with documented stable disease or objective response after at least first line systemic chemotherapy/radiotherapy for advanced disease who have not been treated for the underlying malignant disease for 4 weeks with chemo-, radio- or immunotherapy will be included into the study. The aim of the study is to show safety and tolerability of this immunotherapeutic approach and to investigate efficacy of the immunotherapy.

ELIGIBILITY:
Inclusion Criteria:

* Patients with stage IV metastasized breast or gastric cancer with documented stable disease or objective response after at least first line chemo/ radiotherapy for advanced disease
* HER2 IHC score 2+ on tumor cells, negative FISH result
* HLA-A2 expression
* Female or male patients aged >= 18 years
* Measurable disease according to RECIST criteria
* ECOG 0-1
* Neutrophile count > 1,5x10^9/l
* WBC > 2,5x10^9/l
* Lymphocyte count > 1x10^9/l
* Hemoglobin > 10g/dl
* Platelets > 100x10^9/l
* Normal renal function (creatinine < 150% ULN)
* Normal liver function (Bilirubin < 150% ULN; ALAT/SGPT and ASAT/SGOT < 300% ULN, except proven metastases)
* Expected survival of at least 6 months
* Concomitant anti-hormonal treatment is allowed
* Female patients within child bearing age must have a negative pregnancy test performed not earlier than 21 days before administration of investigational product. Male and female patients with reproductive potential must agree to employ an effective method of birth control throughout the study and for 6 months discontinuation of investigational product. Postmenopausal women must be amenorrheal for at least 12 months to be considered of non-childbearing potential.
* Men and women of childbearing potential must agree to use a highly effective method of birth control which results in a low failure rate (less than 1% per year) when used consistently and correctly.
* Written informed consent that the patient or a legally authorized representative has been informed about all aspects of the study prior to enrollment and is willing to participate and to be included in the study
* Ability to understand and comply with study and follow-up procedures

Exclusion Criteria:

* Treatment with any other investigational drug within 4 weeks prior to the start of the study medication
* Known hypersensitivity to any components of the study product
* Any severe concomitant disease
* Any disease (including psychotic disorders, drug abuse, active infection, uncontrolled hypertension, unstable angina, heart failure, myocardial infarction within the previous year, serious cardiac arrhythmia requiring medication, hepatic, renal or metabolic disease, obstructive or restrictive lung disease) metabolic dysfunction) and physical examination finding likely (in the investigator's opinion) to affect the evaluation of the study or to put patient at risk associated to treatment with the study medication.
* Any heart disease
* Any serious infection or sepsis
* Any autoimmune disorder
* Infection with HIV, chronic infection with Hepatitis B or C
* Any immunodeficiency syndrome
* Surgery within 4 weeks before study entry
* Prior splenectomy
* Brain metastasis or leptomeningeal involvement
* Systemic application of immunosuppressive drugs including systemic corticosteroids within three weeks before study entry
* Patients eligible or treated with any aproved HER2-targeted therapy as Trastuzumab, Pertzuzumab, T-DM1 or Lapatinib
* Radio-, chemo- or immunotherapy other than study medication in parallel or within 4 weeks prior study start
* Active drug abuse or chronic alcoholism
* Pregnancy or breast feeding
* Female and male patients of reproductive potential unwilling or unable to practice a highly effective method of birth control
* History of non-compliance with medical regimens
* Patients unwilling or unable to comply with the protocol

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2014-12; Primary Completion 2017-07-18 (Actual); Study Completion 2018-07-13 (Actual)

PRIMARY OUTCOMES:
Safety and tolerability of HER2-derived peptide vaccination measured by clinical and chemical parameters. | Safety measurement will be assessed up to 113 days relating to start of study treatment
  To examine the safety and tolerability of HER2-derived peptide vaccination in patients with stage IV metastasized breast or gastric cancer with documented stable disease or objective response after at least first line systemic chemotherapy/radiotherapy for advanced disease.

CONTACTS AND LOCATIONS:
Overall Officials: Angela Krackhardt, Prof.Dr.med., Principal Investigator — III.Medizinische Klinik und Poliklinik, Klinikum rechts der Isar der TUM
Locations (1):
- III.Medizinische Klinik und Poliklinik, Klinikum rechts der Isar der TUM, Munich, Bavaria, Germany